CLINICAL TRIAL: NCT00478205
Title: Double-Blind, Parallel-Group Comparison of 23 mg Donepezil Sustained Release (SR) to 10 mg Donepezil Immediate Release (IR) in Patients With Moderate to Severe Alzheimer's Disease
Brief Title: Comparison of 23 mg Donepezil Sustained Release (SR) to 10 mg Donepezil Immediate Release (IR) in Patients With Moderate to Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-G000-326; 2006-004888-54 (EudraCT Number)
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
Keywords: Moderate to Severe Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Aricept (donepezil SR 23 mg)
- 2 (Experimental)
  Interventions: Drug: Aricept (donepezil IR 10 mg)

INTERVENTIONS:
Drug: Aricept (donepezil SR 23 mg) — Patients will receive study medication orally, once daily, for 24 weeks according to a double-dummy design:
  23 mg donepezil SR concurrently with placebo identical in appearance to the 10 mg donepezil IR formulation.
  Other Names: Donepezil hydrochloride
  Arms: 1
Drug: Aricept (donepezil IR 10 mg) — Patients will receive study medication orally, once daily, for 24 weeks according to a double-dummy design:
  10 mg donepezil IR concurrently with placebo identical in appearance to the 23 mg donepezil SR formulation.
  Other Names: Donepezil hydrochloride
  Arms: 2

SUMMARY:
The purpose of this study is to compare 23 mg donepezil sustained release (SR) to the currently marketed formulation of 10 mg donepezil immediate release (IR) in patients with moderate to severe Alzheimer's disease.

DETAILED DESCRIPTION:
This study consists of a double-blind, double-dummy, parallel-group comparison of 23 mg donepezil SR with the currently marketed donepezil formulation (10 mg donepezil IR) in patients with moderate to severe Alzheimer's disease. Patients must have been taking 10 mg IR (or a bioequivalent generic) for at least 3 months prior to Screening. The study will consist of 24 weeks of daily administration of study medication, with clinic visits at Screening, Baseline, 3 weeks (safety only), 6 weeks, 12 weeks, 18 weeks and 24 weeks or early termination. Patients will receive either 10 mg donepezil IR in combination with the placebo corresponding to 23 mg donepezil SR, or 23 mg donepezil SR in combination with the placebo corresponding to 10 mg donepezil IR.

A total of approximately 1600 patients will be enrolled to obtain complete data from approximately 1200 completed patients (Revised per Amendment 02). During the Baseline visit, patients will be randomized in a 2:1 ratio (23 mg donepezil SR to 10 mg donepezil IR). The study will be performed at approximately 200 global sites (Asia, Oceania, Europe, India, Israel, North America, South Africa, and South America) (Revised per Amendments 01 and 02). An Independent Data Monitoring Committee (IDMC) will be established to review safety aspects of the study and to evaluate the results of a planned interim analysis.

Patients who complete the study may be eligible to undergo evaluation for enrollment into the open-label extension study, E2020-G000-328.

ELIGIBILITY:
Inclusion Criteria for Patients:

1. Written informed consent.
2. Patient Age range: Adult patients, 45 to 90 years of age, inclusive.
3. The caregiver must separately meet the specified inclusion/exclusion criteria for caregivers.
4. Women must be of non-child-bearing potential (>1 year post-menopausal or surgically sterile).
5. There must be diagnostic evidence of probable Alzheimer's disease (AD).
6. The patient must have been receiving Aricept at a dose of dose of 10 mg IR (or 10 mg dose of generic donepezil bioequivalent to Aricept), for at least 3 months prior to the Screening visit.
7. A cranial image is required, with no evidence of focal brain disease that would account for dementia.
8. The patient must meet certain psychometric test criteria related to the degree of impairment of cognitive functioning.
9. Health: physically healthy and ambulatory or ambulatory-aided (i.e., walker or cane); corrected vision and hearing sufficient for compliance with testing procedures, and able to read prior to disease onset.
10. Clinical laboratory values must be within normal limits or, if abnormal, must be judged not clinically significant by the investigator.
11. Specified doses of selective serotonin reuptake inhibitors (SSRIs) are allowed in the study if dosage is within approved dose range and stable for 3 months prior to Screening.
12. Other medical conditions, such as hypertension and cardiac disease must be well-controlled and the patient maintained on stable doses of medications for 3 months.
13. Patients with diabetes mellitus or risk factors for diabetes mellitus may be enrolled in the study provided that the patient's disease is stable and that there have been no recent hospitalizations for diabetes complications.
14. Patients whose serum B12 levels at Screening are below the normal range may nonetheless be admitted to the study if they subsequently show normal levels prior to Baseline.
15. Patients with hypothyroidism who are on a stable dose of medication for at least 12 weeks prior to Screening, have normal TSH and free T4 at Screening, and are considered euthyroid will be eligible.
16. Concomitant Medications: Under specified circumstances, the following medications may be allowed: chronic daily benzodiazepine use, bronchodilator medications for treatment of chronic obstructive pulmonary disease (COPD), and memantine. Certain other additional prescription treatments for AD, such as other cholinesterase inhibitors, must have been discontinued for at least 3 months prior to screening.
17. The patient must have a relative/caregiver who supervises the regular taking of the drug at the correct dose and is alert for possible side effects, unless the patient's legal guardian takes on this task.

Inclusion Criteria for Caregivers:

The designated caregiver must be sufficiently familiar with the patient (as determined by the investigator) to provide accurate data. The caregiver must have regular contact with the patient (i.e., an average of 10 or more hours per week), must be able to observe for possible adverse events, and must be able to accompany the patient to all visits.

Exclusion Criteria for Patients:

1. Patients are excluded if they are taking (a) no medication for Alzheimer's disease, (b) Aricept or bioequivalent generic donepezil at doses other than 10 mg daily, or 10 mg for less than 3 months before Screening; (c) other medications for Alzheimer's disease, except that memantine, Vitamin E, fish oil, and/or gingko biloba are allowed if doses have been stable for at least 3 months prior to the Screening visit. Patients undergoing any alternative medical techniques, such as acupuncture or acupressure, specifically for the treatment of AD are not eligible
2. No caregiver available to meet the inclusion criteria for caregivers.
3. Patients who have no measurable blood levels of donepezil in blood samples collected at Screening.
4. Patients with neurological disorders that affect cognition or the ability to assess cognition but are distinguishable from Alzheimer's disease. These include, but are not limited to, Parkinson's disease, multi-infarct dementia, and dementia due to cerebrovascular disease.
5. Patients with psychiatric disorders affecting the ability to assess cognition such as schizophrenia, bipolar or unipolar depression. Patients with clinically significant sleep disorders will also be excluded unless these are controlled by treatment and clinically stable for > 3 months prior to screening.
6. Patients with dementia complicated by other organic disease or Alzheimer's disease with delirium.
7. Patients with drug or alcohol abuse or dependence within the past 5 years according to DSM IV criteria.
8. Patients with any conditions affecting absorption, distribution, or metabolism of the study medication (e.g., inflammatory bowel disease, gastric or duodenal ulcers, hepatic disease, or severe lactose intolerance).
9. Patients with evidence of clinically significant, active gastrointestinal, renal, hepatic, respiratory, endocrine, or cardiovascular system disease (including history of life-threatening arrhythmias).
10. Patients with a history of cancer (does not include basal or squamous cell carcinoma of the skin) treated within 5 years prior to study entry, or current evidence of malignant neoplasm, recurrent, metastatic disease. Males with localized prostate cancer requiring no treatment would not be excluded.
11. Known plan for elective surgery during the treatment period that would require general anesthesia and administration of neuromuscular blocking agents.
12. Donation of blood or blood products during 30 days prior to Screening or plans to donate blood while participating in the study or within 30 days after completion of the study.
13. Patients who are unwilling or unable to fulfill the requirements of the study.
14. Known hypersensitivity to acetylcholinesterase inhibitors or memantine.
15. Use of any prohibited prior or concomitant medications) Any condition that would make the patient, in the opinion of the investigator, unsuitable for the study.
16. Involvement in any other investigational drug clinical trial during the preceding 3 months, or likely involvement in any other such trial during the course of this study.
17. Patients taking concomitant antidepressant medication known to have significant anticholinergic effects, such as tricyclic antidepressants prescribed at doses recommended for the treatment of major depression.
18. Patients who cannot swallow or who have difficult swallowing whole tablets.
19. Patients with fecal and/or urinary incontinence who are unable to cooperate with routine specimen collection.

Exclusion Criteria for Caregivers:

1. Caregivers who are unwilling or unable to give informed consent or otherwise to fulfill the requirements of the study.
2. Caregivers who do not meet certain psychometric test criteria.
3. Any condition that would make the caregiver, in the opinion of the Investigator, unsuitable for the study.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1467 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Yardley, Ph.D, Study Director — Eisai Limted
Locations (1):
- MedTrials, Inc., Hickory, North Carolina, United States

REFERENCES:
- [Derived] Schmitt FA, Saxton J, Ferris SH, Mackell J, Sun Y. Evaluation of an 8-item Severe Impairment Battery (SIB-8) vs. the full SIB in moderate to severe Alzheimer's disease patients participating in a donepezil study. Int J Clin Pract. 2013 Oct;67(10):1050-6. doi: 10.1111/ijcp.12188. PMID 24073978
- [Derived] Salloway S, Mintzer J, Cummings JL, Geldmacher D, Sun Y, Yardley J, Mackell J. Subgroup analysis of US and non-US patients in a global study of high-dose donepezil (23 mg) in moderate and severe Alzheimer's disease. Am J Alzheimers Dis Other Demen. 2012 Sep;27(6):421-32. doi: 10.1177/1533317512454708. PMID 22930699
- [Derived] Doody RS, Geldmacher DS, Farlow MR, Sun Y, Moline M, Mackell J. Efficacy and safety of donepezil 23 mg versus donepezil 10 mg for moderate-to-severe Alzheimer's disease: a subgroup analysis in patients already taking or not taking concomitant memantine. Dement Geriatr Cogn Disord. 2012;33(2-3):164-73. doi: 10.1159/000338236. Epub 2012 May 10. PMID 22572767
- [Derived] Ferris SH, Schmitt FA, Saxton J, Richardson S, Mackell J, Sun Y, Xu Y. Analyzing the impact of 23 mg/day donepezil on language dysfunction in moderate to severe Alzheimer's disease. Alzheimers Res Ther. 2011 Jun 20;3(3):22. doi: 10.1186/alzrt84. PMID 21689411
- [Derived] Farlow M, Veloso F, Moline M, Yardley J, Brand-Schieber E, Bibbiani F, Zou H, Hsu T, Satlin A. Safety and tolerability of donepezil 23 mg in moderate to severe Alzheimer's disease. BMC Neurol. 2011 May 25;11:57. doi: 10.1186/1471-2377-11-57. PMID 21612646
- [Derived] Farlow MR, Salloway S, Tariot PN, Yardley J, Moline ML, Wang Q, Brand-Schieber E, Zou H, Hsu T, Satlin A. Effectiveness and tolerability of high-dose (23 mg/d) versus standard-dose (10 mg/d) donepezil in moderate to severe Alzheimer's disease: A 24-week, randomized, double-blind study. Clin Ther. 2010 Jul;32(7):1234-51. doi: 10.1016/j.clinthera.2010.06.019. PMID 20678673

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil SR 23 mg: Donepezil sustained release (SR) 23 mg in combination with placebo corresponding to donepezil IR 10 mg ; dosing continued for a 24-week treatment period.
- Donepezil IR 10 mg: Donepezil immediate release (IR) 10 mg in combination with placebo corresponding to donepezil SR 23 mg; dosing continued for a 24-week treatment period.
Period: Overall Study
Arm/Group | Donepezil SR 23 mg | Donepezil IR 10 mg
Started | 981 | 486
Completed | 685 | 399
Not Completed | 296 | 87
Not completed — Adverse Event | 182 | 39
Not completed — Medication Non-compliance | 9 | 4
Not completed — Protocol Violation | 15 | 5
Not completed — Request of Investigator or Sponsor | 4 | 5
Not completed — Withdrawal by Subject | 61 | 22
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other | 24 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil SR 23 mg | Donepezil IR 10 mg | Total
Number analyzed (Participants) | 963 | 471 | 1434
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Population
  Years | 73.9 (8.53) | 73.8 (8.56) | 73.8 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population: All patients randomized who took at least one dose of study medication and who had at least one postbaseline safety assessment.
  Participants
    Female | 607 (63.0) | 294 (62.4) | 901 (62.8)
    Male | 356 (37.0) | 177 (37.6) | 533 (37.2)
Race/Ethnicity, Customized [Number; unit: Participants] — Race (Safety Population)
  Participants
    Black | 22 | 9 | 31
    White | 708 | 346 | 1054
    Hispanic | 67 | 26 | 93
    Native American | 0 | 0 | 0
    Asian/Pacific | 161 | 87 | 248
    Other | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in SIB Total Score
Description: The SIB is an assessment of cognitive dysfunction across nine domains such as memory, language, and orientation. The score ranges from 0 (worst) to 100 (best). This outcome was calculated using the LOCF (last observation carried forward) method.
Time Frame: Baseline and Week 24
Population: Intent-to-treat (ITT) population: All Randomized patients in Safety Population and Severe Impairment Battery (SIB) or Clinician Interview-Based Impression of Severity Plus Caregiver Input (CIBIS+) data available at Baseline and SIB or Clinician Interview-Based Impression of Change Plus caregiver Input (CIBIC+ ) data available post-Baseline; LOCF
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Donepezil SR 23 mg | Donepezil IR 10 mg
Number analyzed (Participants) | 909 | 462
Scores on a scale | 2.6 (0.58) | 0.4 (0.66)

2. Secondary Outcome: Change From Baseline to Week 24 in ADCS-ADL Total Score
Description: The ADCS-ADL (Alzhemier's Disease Cooperative Study-Activities of Daily Living) is a 19-item assessment scale used to measure a patient's basic functional abilities, such as walking, grooming, and bathing.Scores range from 0 to 54, with a higher score indicating greater functional ability.
Time Frame: Baseline and Week 24
Population: ITT population, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil SR 23 mg | Donepezil IR 10 mg
Number analyzed (Participants) | 909 | 462
Scores on a scale | -1.2 (6.83) | -1.2 (6.78)

3. Secondary Outcome: Change From Baseline to Week 24 in MMSE Total Score
Description: The MMSE (Mini-Mental State Examination) is a 30-item test that evaluates 5 domains of cognitive function (orientation to time and place, immediate and delayed recall, attention, calculation, and language). The scores range from 0 (most impaired) to 30 (no impaiment).
Time Frame: Baseline and Week 24
Population: ITT population, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil SR 23 mg | Donepezil IR 10 mg
Number analyzed (Participants) | 909 | 462
Scores on a scale | 0.6 (2.93) | 0.4 (3.20)

4. Primary Outcome: Overall Change From Baseline in Modified CIBIC+ to Week 24
Description: The CIBIC+ is a rating scale derived from an interview with the patient and caregiver with an independent rater designed to measure several domains of patient function, such as mental/cognitive state, behavior, and activities of daily living. The scores range from 1 (marked improvement) to 7 (marked worsening).
Time Frame: Baseline and Week 24
Population: ITT population, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil SR 23 mg | Donepezil IR 10 mg
Number analyzed (Participants) | 909 | 462
Scores on a scale | 4.23 (1.07) | 4.29 (1.07)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were recorded from the time of informed consent until after the Final Visit or Early Termination.
Description: Serious adverse events (SAEs) were monitored through the termination visit and through 30 days after study drug discontinuation, whichever was longer.
Arm/Group | Donepezil SR 23 mg | Donepezil IR 10 mg
Serious Adverse Events (participants affected / at risk) | 80/963 | 45/471
Other Adverse Events (participants affected / at risk) | 233/963 | 50/471
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil SR 23 mg (N=963) | Donepezil IR 10 mg (N=471)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1
Bradycardia (Cardiac disorders) | 4 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 2 | 0
Drowning (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 2
Irritability (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 2
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 4 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 5
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 2 | 4
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 3
Delusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Poriomania (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil SR 23 mg (N=963) | Donepezil IR 10 mg (N=471)
Diarrhoea (Gastrointestinal disorders) | 76 | 25
Nausea (Gastrointestinal disorders) | 113 | 16
Vomiting (Gastrointestinal disorders) | 86 | 12
Anorexia (Metabolism and nutrition disorders) | 51 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No